CLINICAL TRIAL: NCT03880747
Title: Incidence of Dumping Syndrome After Laparoscopic Vagus Nerve-preserving Distal Gastrectomy for Early Gastric Cancer
Brief Title: Dumping Syndrome and Quality of Life After Vagus Nerve-preserving Distal Gastrectomy
Acronym: VNP
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBHGS_VNP
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vagus nerve preserving group: Patients who underwent vagus nerve-preserving distal gastrectomy for early gastric cancer
  Interventions: Procedure: Vagus nerve-preserving distal gastrectomy

INTERVENTIONS:
Procedure: Vagus nerve-preserving distal gastrectomy — Laparoscopic distal gastrectomy with the preservation of the celiac and hepatic branch of the vagus nerve.

SUMMARY:
There is no consensus on what type of function-preserving gastrectomy can provide the best patient quality of life (QOL). This study aims to evaluate the incidence of dumping syndrome after vagus nerve-preserving distal gastrectomy (VPNDG).

DETAILED DESCRIPTION:
The study is designed as a prospective observational phase II study with a follow-up period of 12 months. Patients diagnosed with early gastric cancer in the distal 2/3rd of the stomach who are planned to undergo laparoscopic VPNDG with Roux-en Y gastrojejunostomy will be enrolled. Primary endpoint is incidence of dumping syndrome defined by Sigstad score 7 after a 3-month interval. Other outcomes include operative data, early complication, and patient QOL using the European Organization for Research and Treatment of Cancer C-30 and STO22 modules.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with early gastric cancer in the distal 2/3rd of the stomach planned to undergo laparoscopic vagus nerve-preserving distal gastrectomy

Exclusion Criteria:

* Sacrificed vagus nerve
* Anastomosis other than Roux-en Y gastrojejunostomy or uncut Roux-en Y gastrojejunostomy
* conversion to an open procedure
* combined resection of other organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with early gastric cancer in the distal 2/3rd of the stomach
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Dumping syndrome | 1 year
  Sigstad score of equal or more than 7

SECONDARY OUTCOMES:
EORTC C-30/STO22 | 3 months, 6 months, 1 year
  Quality of life surveys
Postoperative complication | 3 months, 6 months, 1 year
  incidence of postoperative complication
Incidence of gallstones | 1 year
  Found in follow-up CT or ultrasound

OTHER OUTCOMES:
Operative time | Immediately after operation
  Time of operation
Estimated blood loss | Immediately after operation
  Blood loss during operation
Time to first flatus | Within 1 week
  Postoperative day to first flatus
Hospital stay | Within 1 week
  Total hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share our IPD with other researchers unless needed.